CLINICAL TRIAL: NCT01782625
Title: Hypercapnia: Cognitive Effects and Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00036937; SPS 181258 (Registry Identifier: Sponsored Programs)
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Hypercapnia; Exercise; Nitrogen Narcosis; Diving; Immersion
Keywords: diving; cognitive impairment; nitrogen narcosis; narcosis; end tidal carbon dioxide; arterial carbon dioxide; immersion
MeSH Terms: conditions — Hypercapnia; Motor Activity; Inert Gas Narcosis; Cognitive Dysfunction; Stupor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- dive to 122 feet, no exercise (Experimental): Subjects will undergo a simulated dive to a maximum depth of 122 feet of seawater with no exercise at depth
  Interventions: Other: NO exercise at depth
- dive to 158 feet, no exercise (Experimental): Subjects will undergo a simulated dive to a maximum depth of 154 feet of seawater with no exercise at depth
  Interventions: Other: NO exercise at depth
- dive to 122 feet, exercise (Experimental): Subjects will undergo a simulated dive to a maximum depth of 122 feet of seawater with exercise at depth
  Interventions: Other: exercise at depth
- dive to 158 feet, exercise (Experimental): Subjects will undergo a simulated dive to a maximum depth of 154 feet of seawater with exercise at depth.
  Interventions: Other: exercise at depth

INTERVENTIONS:
Other: NO exercise at depth — Subjects will NOT exercise while at depth
  Arms: dive to 122 feet, no exercise; dive to 158 feet, no exercise
Other: exercise at depth — Subjects will exercise while at depth
  Arms: dive to 122 feet, exercise; dive to 158 feet, exercise

SUMMARY:
The investigators will simulate the conditions of a working, helmeted diver by using exercising, "head out" immersed subjects to test the following hypotheses:

1. An algorithm can be developed which predicts cognitive performance in immersed exercising divers, based on the exhaled carbon dioxide (PETCO2) and the diver's inspired partial pressures of oxygen and nitrogen (PIO2 and PIN2).
2. PETCO2 using mass spectrometry is an accurate estimate of arterial carbon dioxide (PaCO2) at rest and during immersed exercise and can be used as a PaCO2 surrogate at levels exceeding 50 mmHg and depths up to 158 fsw (gas density 6.4 g/l, similar to 165 fsw density of 6.8 g/l).

ELIGIBILITY:
Inclusion Criteria:

* healthy,
* male,
* age greater than 18,
* age less than 50

Exclusion Criteria:

* smoker,
* asthma,
* cardiac disease,
* inability to pedal a bicycle ergometer,
* inability to perform vigorous exercise

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Is cognitive ability different while resting versus compared to cognitive ability while diving, breathing different gas mixtures and while exercising? | pre-dive to dive to post-dive (approximately 2 hours)
  Subjects will undergo computerized cognitive testing before, during and after a simulated dive in the Duke Hyperbaric Chamber. Different exercise conditions (rest or exercise) and different breathing gas mixtures (added carbon dioxide or not)will be assessed and compared to the pre-dive conditions.

SECONDARY OUTCOMES:
How does exhaled (end tidal) carbon dioxide compare with arterial carbon dioxide? | pre-dive to dive to post dive (approximately 2 hours)
  Exhaled (end tidal) carbon dioxide will be compared to arterial carbon dioxide at the various experimental conditions of the study (at the surface versus during the dive, during exercise versus during rest, breathing gas with added carbon dioxide versus breathing gas without added carbon dioxide)

CONTACTS AND LOCATIONS:
Overall Officials: John J Freiberger, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Hyperbaric Medicine and Environmental Physiology, Durham, North Carolina, United States